CLINICAL TRIAL: NCT06690554
Title: The Effect of Education Given to Preconception Women in Line with the Health Promotion Model on Fertility Awareness, Preconception Knowledge and Attitude Levels
Brief Title: Health Promotion Model, Fertility Awareness, Preconception Knowledge and Attitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/1011
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-11

CONDITIONS: Fertility Issues; Preconception Injuries; Health Behavior
Keywords: Fertility Awareness; Preconceptional Knowledge and Attitude; Health Promotion Model
MeSH Terms: conditions — Infertility; Preconception Injuries; Health Behavior; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (No Intervention): * Information about the research will be provided.
  * Written consent will be obtained.
  * Personal Information Form, Fertility Awareness, Preconceptional Knowledge and Attitude will be applied to women who accept to participate in the research.
  * Five days after the first interview, women will be reached and the scales will be applied.
  * Three months after the first interview, women will be reached, invited to the institution and the scales will be applied again.
- Education Group (Experimental): Women will be given a five-day training in line with the health promotion model.
  * Information will be provided to women who apply to the hospital.
  * Written consent documents will be obtained from women who agree to participate in the study.
  * Women assigned to the intervention group will attend classes in groups of 8-10.
  * Women will be given a 60-minute training once a day for five days.
  * The total training duration is five hours.
  * Scales will be applied to women who complete the training at the end of the fifth day.
  * Women who have completed the training will be contacted by phone at the end of the first and second months, reminded of health promotion behaviors and their questions will be answered and follow-ups will be carried out.
  * At the end of the third month, women who have received training will be invited to the institution and the Fertility Awareness, Preconceptional Knowledge and Attitude will be filled out face-to-face for the final test.
  Interventions: Other: Education Group

INTERVENTIONS:
Other: Education Group — Women will be given a five-day training in line with the health promotion model.
  Information will be provided to women who apply to the hospital. Written consent documents will be obtained from women who agree to participate in the study.
  Women assigned to the intervention group will attend classes in groups of 8-10. Women will be given a 60-minute training once a day for five days. The total training duration is five hours. Scales will be applied to women who complete the training at the end of the fifth day.
  Women who have completed the training will be contacted by phone at the end of the first and second months, reminded of health promotion behaviors and their questions will be answered and follow-ups will be carried out.
  At the end of the third month, women who have received training will be invited to the institution and the Fertility Awareness, Preconceptional Knowledge and Attitude will be filled out face-to-face for the final test.
  Arms: Education Group

SUMMARY:
The effect of education given to preconceptional women in line with the health promotion model on fertility awareness, preconceptional knowledge and attitude levels

DETAILED DESCRIPTION:
The research is a randomized controlled trial. The research will conducted with 128 women (intervention group n=64, control group n=64). It will consist of women between the ages of 18-35 who applied to the community health unit of Güneysınır District Health Directorate between December 2024-May 2025.

Women who accept the research and are assigned to the intervention group will be given a five-day training to increase fertility awareness and preconceptional knowledge levels in line with the health promotion model. At the end of the fifth day, the Fertility Awareness Scale, Preconceptional Knowledge and Attitude Scale, and the Clinical Evaluation Form of the Health Promotion Plan for the Health Promotion Model will be applied to women who complete the training with a face-to-face interview technique. The women in the intervention group will be reached by phone at the end of the first and second months to remind them of their health promotion behaviors and to answer their questions and carry out follow-ups. At the end of the third month, women who have completed the training will be invited to the institution and the forms will be filled out again.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-35,
* Planning to get pregnant within a year,
* Literate,
* Can understand and speak Turkish,
* Agree to participate in the research.

Exclusion Criteria:

* Women who are pregnant,
* Women who are breastfeeding,
* Women who have been diagnosed with infertility,
* Women who have a history of chronic disease (hypertension, diabetes mellitus, hypothyroidism, etc.),
* Women who have a sexually transmitted disease (HIV, HPV, etc.),
* Women who have a physical disability,
* Women who have a psychiatric disease,
* Women who have a history of gynecological disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of sociodemographic of women | 4 months
  Sociodemographic of women will be collected through surveys and compared and reported
Comparison of obstetric features of women | 4 months
  Obstetric features of women will be collected through surveys and compared and reported
Comparison of women's fertility awareness scale average scores by groups | 4 months
  The fertility awareness scale will be applied to women. The fertility awareness scale is 19-95 points (min-max), and as the score increases, fertility awareness scale increases.
Comparison of women's preconceptional knowledge and attitude scale average scores by groups | 4 months
  Preconceptional knowledge and attitude scale will be applied to women. The preconceptional knowledge and attitude scaleis 43-215 points (min-max), and as the score increases, preconceptional knowledge and attitude increases.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çankaya, Principal Investigator — Selcuk University
Locations (1):
- Seyhan Çankaya, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No